CLINICAL TRIAL: NCT02499211
Title: The Impact of Healthy Food Marketing Strategies in Supermarkets
Brief Title: Healthy In-Store Marketing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Principal Investigator, Karen Glanz, George A Weiss University Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 820635
Record Dates: First submitted 2015-06-30; First posted 2015-07-16 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: obesity; health disparities; healthy food marketing; food environments; marketing environments; food access; food purchase decision making
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention stores (Experimental): Supermarkets will be the unit of randomization, intervention, and analysis. During randomization, stores are paired by size and percent sales of Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) and Supplemental Nutrition Assistance Program (SNAP) funding. The intervention will last for 2 years, and will consist of in-store marketing of healthier (lower calorie) products through placement and promotion strategies in 6 food and beverage categories: milk; frozen meals; beverages in checkout coolers; bread; salty snacks; and cheese.
  Interventions: Other: Intervention stores
- Non-intervention stores (No Intervention): No intervention administered. Supermarkets will be the unit of randomization, intervention, and analysis. During randomization, stores are paired by size and percent sales of WIC and SNAP funding. The non-intervention stores will not receive an intervention.

INTERVENTIONS:
Other: Intervention stores — In-store marketing strategies will focus on placement and promotion of healthier items (lower calorie options) in the milk, frozen food, beverage checkout cooler, bread, salty snacks, and cheese sections of the store.
  Intervention efforts in the dairy section promote lower calorie milk (skim, 1%, and 2%), while diminishing the presence of whole milk. The visual order of the milk displays will be changed, and the number of facings, or the fronts of packages the consumer can see, of whole milk will be decreased by 30% while increasing the facings of the lower calorie milk. In the other product categories, target products will be moved to eye level and the number of facings will be increased.
  Call-out signs will be placed by the target products that list the name and price of the product. No health information or claims will be included. Signage will be rotated monthly to increase the chances that customers will notice them.
  Arms: Intervention stores

SUMMARY:
Using a cluster randomized controlled design, this study will evaluate effects of in-store healthy food marketing strategies on sales and purchase of specific healthier items in six product categories (milk, frozen entrees, beverage checkout coolers, salty snacks, bread and cheese); and examine the effects of changes in in-store food marketing environments on sales of healthier foods. If these strategies are found to be effective, they could be used widely to encourage healthy retail sales, complement food access initiatives, and reduce health disparities in obesity and other diseases. Supermarkets will be the unit of randomization, intervention, and analysis.

DETAILED DESCRIPTION:
As the prevalence of obesity has increased, public health experts have increasingly focused on the environments that shape overeating and unhealthy food choices. Retail grocery stores are pivotally positioned to influence choices and favorably affect energy balance. Greater availability of healthier foods, if translated to health-promoting purchases, can positively affect diet quality among those at greatest risk for obesity- low-income, ethnic minorities.

The aims of the proposed study are:

1. To evaluate, in a cluster randomized controlled trial design, effects of in-store healthy food marketing strategies on sales and purchase of healthier items in six product categories (milk, frozen entrees, beverage checkout coolers, bread, salty snacks and cheese); and
2. To evaluate the association of changes in supermarket food marketing environments with changes in sales of specific healthier food items in the same six product categories; and
3. To examine the relationships between neighborhood characteristics and changes in sales and purchases of healthier items in the six product categories.

Investigators hypothesize that sales of targeted products will be significantly higher, and that more health-focused food marketing environments will be associated with higher sales of healthy food items.

The study will be conducted in 32 supermarkets in urban, low-income, high-minority neighbor-hoods in the mid-Atlantic and Northeast regions. Intervention strategies will include prime placement, increased visibility of healthier products, call-out signs, and taste-testing for milk. Control stores will be assessment-only. Supermarket chains will help implement the strategies and provide data on sales of targeted products. Interventions will be conducted for 2 years, with an emphasis on scalability and long-term sustainability. The primary outcome measures of purchasing will be weekly sales per store for each product. Individual purchasing will be assessed in a cohort of shoppers by interviews and shopping receipts. The Grocery Marketing Environment Assessment (GMEA) tool will be used to assess marketing environments.

The research team completed a randomized pilot study of a 6-month intervention in eight supermarkets, which demonstrated the impact of the interventions on three food categories. The proposed study will provide an expanded and extended, larger-scale, rigorous test of novel and widely applicable strategies to encourage healthy retail sales, complement increased-access initiatives, and reduce health disparities in obesity and related diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Do most of your food shopping at the store where they are recruited
* Speak English
* Be the main household shopper

Exclusion Criteria:

* No exclusion criteria defined

  * Eligible stores will be at least 35,000 square feet in size, and be located in urban or suburban communities with at least 50% of households below the state median income.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Weekly sales data by units sold | up to 36 months
  Store IT managers will provide weekly sales data for the targeted products. The data will include units sold of all targeted products (higher calorie versions and lower-calorie alternatives).

SECONDARY OUTCOMES:
Marketing environment in the grocery stores using GMEA | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  Observations will examine the food promotion environment in supermarkets, including the presence of promotional displays. Summary scores of the amount and visibility of product promotions will be computed for each target product, for other measured products (e.g., produce, cereal), and for the store as a whole using the Grocery Marketing Environment Assessment (GMEA) tool.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Foster GD, Karpyn A, Wojtanowski AC, Davis E, Weiss S, Brensinger C, Tierney A, Guo W, Brown J, Spross C, Leuchten D, Burns PJ, Glanz K. Placement and promotion strategies to increase sales of healthier products in supermarkets in low-income, ethnically diverse neighborhoods: a randomized controlled trial. Am J Clin Nutr. 2014 Jun;99(6):1359-68. doi: 10.3945/ajcn.113.075572. Epub 2014 Apr 2. PMID 24695894